CLINICAL TRIAL: NCT05530239
Title: Single-center Pilot Study: Nano-rheological Biomarkers for Patients With Sickle Cell Disease (SCD) Versus Control Subjects (Other Constitutional Red Blood Cell Diseases and Healthy Subjects)
Brief Title: Nano-rheological Biomarkers for Patients With Sickle Cell Disease (SCD) Versus Control Subjects (Other Constitutional Red Blood Cell Diseases and Healthy Subjects)
Acronym: DREPNANO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0135
Record Dates: First submitted 2022-07-25; First posted 2022-09-07 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-07

CONDITIONS: Sickle Cell Disease
Keywords: Hemorheology; Microfluidics; Blood viscosity; Red blood cell; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects: Subjects with no documented hematological pathology (neither constitutional nor acquired). From the recruitment of living kidney donors, transplantation unit of Grenoble Alpes University Hospital
  Interventions: Other: Blood sample collection
- SCD patients: Patients with SCD
  Interventions: Other: Blood sample collection
- Control patients: With a constitutional non-sickle cell disease of the red blood cell, or an acquired red blood cell disease.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection

SUMMARY:
Numerous pathologies (sickle cell disease, thalassemia, spherocytosis, etc.) lead to changes in the rheological properties of the blood, in particular via alterations in the deformability of red blood cells. These alterations lead to circulatory complications of which an emblematic example is the sickle cell crisis which manifests itself by microcirculatory occlusions. Several authors suggest that the deformability of erythrocytes is a key parameter for the diagnosis and monitoring of patients. Numerous studies, especially in vitro, show that the mechanical properties of the red blood cell significantly influence its dynamics in flow (blood viscosity, distribution in capillary networks). Moreover, concerning the specific problem of vaso-occlusion, the proportion of the most rigid red blood cells is a determining factor of the probability of occlusion more than the average value of this rigidity which can hide great disparities.

There is no clinically usable test to assess the alteration of the fine rheology of the red blood cell in a patient. Functional tests such as ektacytometry require heavy equipment and teams of specialized biologists; this technique is therefore only available in 3 biological reference centers in France. "Mechanical phenotyping" seems to be a potentially simpler and more accessible technique, and has already shown promising prospects in other nosological settings than red blood cell pathologies.

Today, there is no specific marker of sickle cell vaso-occlusive crisis, nor marker of severity, that would be useful for pathophysiological understanding but also for clinical management.

DETAILED DESCRIPTION:
This study aims to characterize the microfluidic flow and intra-erythrocyte viscosity of sickle cell red blood cells, and to identify specific biological phenotype or clinical severity profiles. The techniques used are microfluidic circuits for the study of flow and molecular rotors for the measurement of intra-erythrocyte viscosity, using deoxygenation cycles in order to model physio-pathological situations.

The first part will allow the calibration of the microfluidic techniques used (microfluidic circuit and molecular rotors), testing blood from healthy subjects (without constitutional or acquired red blood cell pathology) and blood from SCD patients. The aim is to define the reproducibility and sensitivity of the techniques.

A second part is aimed at establishing a rheological profile of the blood of patients with SCD in comparison with blood from control subjects, i.e. with other constitutional or acquired red blood cell pathology.

ELIGIBILITY:
Inclusion Criteria for healthy volunteers :

1. Patient age ≥ 18 years
2. With social care protection
3. Living donor recruited for kidney donation with normal blood count

Inclusion Criteria for SDC patient :

1. Patient age ≥ 18 years
2. With social care protection
3. SCD patient with documented phenotype: SS, S°, S+, SC, SLepore, SOrab, SDPundjab, ASantilles... with or without specific treatment

Inclusion Criteria for patient with a constitutional non-sickle cell disease of the red blood cell, or an acquired red blood cell disease :

1. Patient age ≥ 18 years
2. With social care protection
3. With any of the following conditions :

   1. Patient being managed for anemia due to martial deficiency, and prior to oral or intravenous replacement therapy
   2. Patient being followed for myeloproliferative syndrome at diagnosis, and prior to any specific treatment (hemodilution or hydroxycarbamide or other specific treatment)
   3. A patient with a MCGRE other than a major sickle cell syndrome, whether or not under specific treatment
   4. Hemoglobinopathy: transfusion-dependent or independent thalassemias (major or intermediate), thalassemias minor, heterozygous sickle cell trait A/S, other heterozygous hemoglobin variants (C, E, Lepore...), hyperaffine hemoglobin
   5. Membrane disorders (hereditary spherocytosis)
   6. Canalopathies (stomatocytosis with dehydrated or hyperhydrated erythrocytes, melanesian ovalocytosis...)
   7. Enzyme deficiencies (G6PD, PK, GPI...)

Exclusion Criteria for all patients:

1. Patient age < 18 years
2. Subject under guardianship, or subject deprived of freedom
3. Linguistic or literacy status not allowing for informed consent despite patient information in "Easy to Read and Understand" format
4. Known history of HIV, HTLV, syphilis, or positive serology and active viral hepatitis B or C.

   Additional Exclusion Criteria for healthy volunteers :
5. Abnormal blood count, or possible martial deficiency with ferritin levels below 50µg/l, or current treatment with hydroxycarbamide, or transfusion within 4 months prior to inclusion.

Additional Exclusion Criteria for SCD patient :

5) Treatment with hydroxycarbamide started less than 6 months ago 6) Anemia with hemoglobin level <60g/l in the absence of cardiorespiratory pathology, <70g/l in pregnancy, or in the presence of cardiorespiratory pathology that may alter the tolerance of anemia.

Additional Exclusion Criteria for patient with a constitutional non-sickle cell disease of the red blood cell, or an acquired red blood cell disease :

5) Anemia with hemoglobin level <60g/l, <70g/l in pregnancy, or in the presence of cardio-respiratory pathology that may alter the tolerance of anemia.

6) Diagnosis not finalized (in progress), or uncertain nosological framework, or diagnostic wandering.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be patient with sickle cell disease (SCD) in comparaison of two populations : healthy volunteers (living donor of kidney) and patient with a constitutional non-sickle cell disease of the red blood cell, or an acquired red blood cell disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Study of the intra-erythrocyte viscosity dispersion and rheological profile of red blood cells | 30 months
  Measure of the intra-erythrocyte viscosity dispersion using molecular rotors technique, study of rheological profile of red blood cells in microfluidic circuit : measure of the speed of flowing, and DI deformability Index [DI = (L-W)/(L+W)] of each red blood cell, DI dispersion in each sample, in basal state and after exposure to deoxygenation cycles of blood SCD patients versus control subjects.

SECONDARY OUTCOMES:
Study of the intra-erythrocyte viscosity dispersion and rheological profile of red blood cells | 24 months
  Measure of the intra-erythrocyte viscosity dispersion using molecular rotors technique, study of rheological profile of red blood cells in microfluidic circuit : measure of the speed of flowing, and DI deformability Index [DI = (L-W)/(L+W)] of each red blood cell, DI dispersion in each sample, in basal state and after exposure to deoxygenation cycles in different conditions : congenital red blood cell disorders, acquired red blood cell disorders and clinical events (vasoocclusive crisis, pregnancy, infection).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MAKOWSKI, mD, Principal Investigator — CHU Grenoble Alpes

REFERENCES:
- [Background] Arlet JB. [A new therapeutic era in sickle cell disease]. Rev Med Interne. 2017 Sep;38(9):569-571. doi: 10.1016/j.revmed.2017.05.006. Epub 2017 Jun 16. No abstract available. French. PMID 28624233
- [Background] Ataga KI, Kutlar A, Kanter J. Crizanlizumab in Sickle Cell Disease. N Engl J Med. 2017 May 4;376(18):1796. doi: 10.1056/NEJMc1703162. No abstract available. PMID 28467874
- [Background] Ballas SK, Barton FB, Waclawiw MA, Swerdlow P, Eckman JR, Pegelow CH, Koshy M, Barton BA, Bonds DR. Hydroxyurea and sickle cell anemia: effect on quality of life. Health Qual Life Outcomes. 2006 Aug 31;4:59. doi: 10.1186/1477-7525-4-59. PMID 16942629
- [Background] Ballas SK. The Evolving Pharmacotherapeutic Landscape for the Treatment of Sickle Cell Disease. Mediterr J Hematol Infect Dis. 2020 Jan 1;12(1):e2020010. doi: 10.4084/MJHID.2020.010. eCollection 2020. PMID 31934320
- [Background] Baez S, Kaul DK, Nagel RL. Microvascular determinants of blood flow behavior and HbSS erythrocyte plugging in microcirculation. Blood Cells. 1982;8(1):127-37. No abstract available. PMID 7115970
- [Background] Banerjee R, Nageshwari K, Puniyani RR. The diagnostic relevance of red cell rigidity. Clin Hemorheol Microcirc. 1998 Sep;19(1):21-4. PMID 9806729
- [Background] Bartolucci P, Brugnara C, Teixeira-Pinto A, Pissard S, Moradkhani K, Jouault H, Galacteros F. Erythrocyte density in sickle cell syndromes is associated with specific clinical manifestations and hemolysis. Blood. 2012 Oct 11;120(15):3136-41. doi: 10.1182/blood-2012-04-424184. Epub 2012 Aug 23. PMID 22919030
- [Background] Briole A, Podgorski T, Abou B. Molecular rotors as intracellular probes of red blood cell stiffness. Soft Matter. 2021 May 5;17(17):4525-4537. doi: 10.1039/d1sm00321f. PMID 33949619
- [Background] Connes P, Alexy T, Detterich J, Romana M, Hardy-Dessources MD, Ballas SK. The role of blood rheology in sickle cell disease. Blood Rev. 2016 Mar;30(2):111-8. doi: 10.1016/j.blre.2015.08.005. Epub 2015 Aug 28. PMID 26341565
- [Background] Du E, Diez-Silva M, Kato GJ, Dao M, Suresh S. Kinetics of sickle cell biorheology and implications for painful vasoocclusive crisis. Proc Natl Acad Sci U S A. 2015 Feb 3;112(5):1422-7. doi: 10.1073/pnas.1424111112. Epub 2015 Jan 20. PMID 25605910
- [Background] Faivre M, Renoux C, Bessaa A, Da Costa L, Joly P, Gauthier A, Connes P. Mechanical Signature of Red Blood Cells Flowing Out of a Microfluidic Constriction Is Impacted by Membrane Elasticity, Cell Surface-to-Volume Ratio and Diseases. Front Physiol. 2020 Jun 12;11:576. doi: 10.3389/fphys.2020.00576. eCollection 2020. PMID 32595519
- [Background] Gladwin MT, Vichinsky E. Pulmonary complications of sickle cell disease. N Engl J Med. 2008 Nov 20;359(21):2254-65. doi: 10.1056/NEJMra0804411. No abstract available. PMID 19020327
- [Background] Guo Q, Duffy SP, Matthews K, Santoso AT, Scott MD, Ma H. Microfluidic analysis of red blood cell deformability. J Biomech. 2014 Jun 3;47(8):1767-76. doi: 10.1016/j.jbiomech.2014.03.038. Epub 2014 Apr 5. PMID 24767871
- [Background] Gossett DR, Tse HT, Lee SA, Ying Y, Lindgren AG, Yang OO, Rao J, Clark AT, Di Carlo D. Hydrodynamic stretching of single cells for large population mechanical phenotyping. Proc Natl Acad Sci U S A. 2012 May 15;109(20):7630-5. doi: 10.1073/pnas.1200107109. Epub 2012 Apr 30. PMID 22547795
- [Background] Hamideh D, Alvarez O. Sickle cell disease related mortality in the United States (1999-2009). Pediatr Blood Cancer. 2013 Sep;60(9):1482-6. doi: 10.1002/pbc.24557. Epub 2013 Apr 23. PMID 23637037
- [Background] Holmes D, Whyte G, Bailey J, Vergara-Irigaray N, Ekpenyong A, Guck J, Duke T. Separation of blood cells with differing deformability using deterministic lateral displacement(dagger). Interface Focus. 2014 Dec 6;4(6):20140011. doi: 10.1098/rsfs.2014.0011. PMID 25485078
- [Background] Kaul DK, Fabry ME, Windisch P, Baez S, Nagel RL. Erythrocytes in sickle cell anemia are heterogeneous in their rheological and hemodynamic characteristics. J Clin Invest. 1983 Jul;72(1):22-31. doi: 10.1172/jci110960. PMID 6874947
- [Background] Kaul DK, Fabry ME. In vivo studies of sickle red blood cells. Microcirculation. 2004 Mar;11(2):153-65. PMID 15280089
- [Background] Kuimova MK, Yahioglu G, Levitt JA, Suhling K. Molecular rotor measures viscosity of live cells via fluorescence lifetime imaging. J Am Chem Soc. 2008 May 28;130(21):6672-3. doi: 10.1021/ja800570d. Epub 2008 May 6. PMID 18457396
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. Mortality rates and age at death from sickle cell disease: U.S., 1979-2005. Public Health Rep. 2013 Mar-Apr;128(2):110-6. doi: 10.1177/003335491312800206. PMID 23450875
- [Background] Lipowsky HH, Cram LE, Justice W, Eppihimer MJ. Effect of erythrocyte deformability on in vivo red cell transit time and hematocrit and their correlation with in vitro filterability. Microvasc Res. 1993 Jul;46(1):43-64. doi: 10.1006/mvre.1993.1034. PMID 8412852
- [Background] Lu X, Chaudhury A, Higgins JM, Wood DK. Oxygen-dependent flow of sickle trait blood as an in vitro therapeutic benchmark for sickle cell disease treatments. Am J Hematol. 2018 Oct;93(10):1227-1235. doi: 10.1002/ajh.25227. Epub 2018 Aug 21. PMID 30033564
- [Background] Niihara Y, Miller ST, Kanter J, Lanzkron S, Smith WR, Hsu LL, Gordeuk VR, Viswanathan K, Sarnaik S, Osunkwo I, Guillaume E, Sadanandan S, Sieger L, Lasky JL, Panosyan EH, Blake OA, New TN, Bellevue R, Tran LT, Razon RL, Stark CW, Neumayr LD, Vichinsky EP; Investigators of the Phase 3 Trial of l-Glutamine in Sickle Cell Disease. A Phase 3 Trial of l-Glutamine in Sickle Cell Disease. N Engl J Med. 2018 Jul 19;379(3):226-235. doi: 10.1056/NEJMoa1715971. PMID 30021096
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290
- [Background] Ribeil JA, Hacein-Bey-Abina S, Payen E, Magnani A, Semeraro M, Magrin E, Caccavelli L, Neven B, Bourget P, El Nemer W, Bartolucci P, Weber L, Puy H, Meritet JF, Grevent D, Beuzard Y, Chretien S, Lefebvre T, Ross RW, Negre O, Veres G, Sandler L, Soni S, de Montalembert M, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in a Patient with Sickle Cell Disease. N Engl J Med. 2017 Mar 2;376(9):848-855. doi: 10.1056/NEJMoa1609677. PMID 28249145
- [Background] Tomaiuolo G. Biomechanical properties of red blood cells in health and disease towards microfluidics. Biomicrofluidics. 2014 Sep 17;8(5):051501. doi: 10.1063/1.4895755. eCollection 2014 Sep. PMID 25332724
- [Background] Telen MJ. Developing new pharmacotherapeutic approaches to treating sickle-cell disease. ISBT Sci Ser. 2017 Feb;12(1):239-247. doi: 10.1111/voxs.12305. Epub 2016 Nov 15. PMID 28484512
- [Background] Vargas FF, Blackshear GL. Vascular resistance and transit time of sickle red blood cells. Blood Cells. 1982;8(1):139-45. PMID 7115971
- [Background] Woodcock EM, Girvan P, Eckert J, Lopez-Duarte I, Kubankova M, van Loon JJWA, Brooks NJ, Kuimova MK. Measuring Intracellular Viscosity in Conditions of Hypergravity. Biophys J. 2019 May 21;116(10):1984-1993. doi: 10.1016/j.bpj.2019.03.038. Epub 2019 Apr 8. PMID 31053255
- [Background] Yaginuma T, Oliveira MS, Lima R, Ishikawa T, Yamaguchi T. Human red blood cell behavior under homogeneous extensional flow in a hyperbolic-shaped microchannel. Biomicrofluidics. 2013 Sep 24;7(5):54110. doi: 10.1063/1.4820414. eCollection 2013. PMID 24404073